CLINICAL TRIAL: NCT03061045
Title: Contrast Enhanced Ultrasound Evaluation of Brain Perfusion in Neonatal Post-Hemorrhagic Hydrocephalus
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI is leaving the institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00129090
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Neonatal Post-Hemorrhagic Hydrocephalus
MeSH Terms: interventions — Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contrast Enhanced Brain Ultrasound (Experimental): Neonates with post-hemorrhagic hydrocephalus recruited for this study will all undergo contrast enhanced ultrasound examination of the head, a diagnostic intervention for the study.
  Interventions: Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 MG Intravenous Powder for Suspension [LUMASON]

INTERVENTIONS:
Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 MG Intravenous Powder for Suspension [LUMASON] — All patients enrolled in this study will undergo contrast enhanced ultrasound examination for assessment of brain perfusion.

SUMMARY:
The aim of the proposed project is therefore to utilize the CEUS technique to assess cerebral perfusion changes before and after ventricular shunting in neonatal cases of PHH. The expectation of the proposed project is to validate statistically significant cerebral perfusion differences before and after shunting in neonates with PHH, as a preliminary feasibility study prior to conducting a large scale, prospective clinical trial incorporating therapeutic interventions using the CEUS technique.

DETAILED DESCRIPTION:
Timely decompression of post-hemorrhagic hydrocephalus (PHH) due to intraventricular hemorrhage in premature babies is key to reducing long-term cognitive and motor disability. Exactly when to place a ventricular shunt for decompression and alleviation of increased intracranial pressure (ICP) remains a dilemma for neurosurgeons, and the only guidance is based on changes in size of the ventricles not necessarily reflective of cerebral hemodynamics. There is a dire need for a novel diagnostic tool that can perform serial, bedside assessment of cerebral perfusion. At times, intermittent shunting may be needed depending on the dynamic changes in brain perfusion, and this is not practical with the current diagnostic tools. While most diagnostic techniques require sedation or transport (i.e. magnetic resonance imaging), few available bedside techniques (i.e. near infrared spectroscopy or Doppler ultrasound) are limited soft tissue contrast, depth of penetration, and/or ability to quantify cerebral perfusion. Potential long-term effects of sedation in neonates are also relatively unknown. In this regard, contrast enhanced ultrasound (CEUS) is easily repeatable technique that can be performed at bedside in less than 5 minutes and provide dynamic cerebral perfusion quantification. The aim of the proposed project is therefore to utilize the CEUS technique to detect cerebral perfusion changes before and after ventricular shunting in neonatal cases of PHH. The specific hypothesis behind the proposed research is that impaired cerebral perfusion in PHH correlates with long-term cognitive and motor disability. The hypothesis is based on the following evidence. First, substantial data from animal studies of hydrocephalus demonstrate a significant role of impaired cerebral hemodynamics in the pathophysiology of brain injury in PHH. Second, animal studies have clearly shown that early treatment of hydrocephalus reduces brain injury and cognitive development. Third, preliminary studies of human infants validate aforementioned findings from animal studies. The expectation of the proposed project is to validate statistically significant cerebral perfusion differences before and after shunting in neonates with PHH, as a preliminary feasibility study prior to conducting a large scale, prospective clinical trial incorporating therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Preexisting IV line
* Stable clinical condition
* No prior allergy to ultrasound contrast agents
* Presence of post-hemorrhagic hydrocephalus

Exclusion Criteria:

* Unstable clinical condition
* Inability to complete the exam
* Allergy to ultrasound contrast agents

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Wash-In Slope (Intensity in dB/Sec) | Immediately before and after ventricular shunting
  Wash-In Slope as derived from contrast enhanced ultrasound perfusion kinetics curve will be obtained as one quantifiable measure of brain perfusion in neonates with post-hemorrhagic hydrocephalus.
Peak Intensity (Intensity in dB) | Immediately before and after ventricular shunting
  Peak Intensity as derived from contrast enhanced ultrasound perfusion kinetics curve will be obtained as one quantifiable measure of brain perfusion in neonates with post-hemorrhagic hydrocephalus.
Time to Peak (sec) | Immediately before and after ventricular shunting
  Time to Peak as derived from contrast enhanced ultrasound perfusion kinetics curve will be obtained as one quantifiable measure of brain perfusion in neonates with post-hemorrhagic hydrocephalus.
Area Under the Curve (Intensity in dB x sec) | Immediately before and after ventricular shunting
  Area Under the Curve as derived from contrast enhanced ultrasound perfusion kinetics curve will be obtained as one quantifiable measure of brain perfusion in neonates with post-hemorrhagic hydrocephalus.
Mean Transit Time (sec) | Immediately before and after ventricular shunting
  Mean Transit Time as derived from contrast enhanced ultrasound perfusion kinetics curve will be obtained as one quantifiable measure of brain perfusion in neonates with post-hemorrhagic hydrocephalus.
Time to Peak to 1/2 (sec) | Immediately before and after ventricular shunting
  Time to peak to 1/2 as derived from contrast enhanced ultrasound perfusion kinetics curve will be obtained as one quantifiable measure of brain perfusion in neonates with post-hemorrhagic hydrocephalus.

CONTACTS AND LOCATIONS:
Overall Officials: Misun Hwang, M.D., Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No